CLINICAL TRIAL: NCT04581577
Title: Perceptions of the Clinical and Psychosocial Impact of Covid-19 in Patients With Neuromuscular and Neurological Disorders
Brief Title: Perceptions of the Clinical and Psychosocial Impact of Covid-19 in Patients With NMD
Acronym: CLASSIC
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 286495
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Neuromuscular Diseases; Neurological Diseases or Conditions
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult patients with neuromuscular or neurological disorders: Telephone questionnaires administered directly to patients over 16 years of age with neuromuscular or neurological disorders
  Interventions: Other: Semi-structured telephone questionnaire
- Parents of paediatric patients with neuromuscular or neurological disorders: Telephone questionnaires administered to the parents of patients over 16 years of age with neuromuscular or neurological disorders
  Interventions: Other: Semi-structured telephone questionnaire

INTERVENTIONS:
Other: Semi-structured telephone questionnaire — Semi-structured telephone questionnaire

SUMMARY:
This study aims to evaluate perceived clinical and psychosocial experiences of patients and their families during the Covid-19 pandemic. it is important to understand the implications of the pandemic for this population, particularly given its likely protracted course, and resultant limitations to daily activities and clinical care. This will help clinicians plan support and adaptations to the services they provide in the medium to long term.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

Adult group

* Patient over 16 years of age with a confirmed diagnosis of neuromuscular and/or neurological disorder
* Able and willing to provide informed consent

Paediatric group

* Parent of a patient under 16 years of age with a confirmed diagnosis of neuromuscular and/or neurological disorder
* Able and willing to provide informed consent

Exclusion Criteria:

* Unwilling for telephone questionnaire to be audio-recorded

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of a neuromuscular and/or neurological disorder including Duchenne muscular dystrophy, spinal muscular atrophy, congenital muscular dystrophies, and other neuromuscular and neurological disorders
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Qualitative evaluation of the perceived clinical and psychosocial impact of the Covid-19 pandemic in patients with neuromuscular and neurological disorders | 4 months
  Evaluation of semi-structured questionnaires using thematic analysis

SECONDARY OUTCOMES:
Quantification of the proportion of patients with NMD who have had suspected or confirmed Covid-19 infection during the pandemic | 4 months
  Quantitative analysis of the proportion of questionnaire respondents reporting confirmed or suspected Covid-19 infection
Qualitative evaluation of the social environment of patients with NMDs | 4 months
  Qualitative analysis describing the social environment of patients with NMDs
Qualitative evaluation of the social activities of patients with NMDs | 4 months
  Qualitative analysis describing the social activities of patients with NMDs
Qualitative evaluation of the professional activities of patients with NMDs | 4 months
  Qualitative analysis describing the professional activities of patients with NMDs
Qualitative evaluation of the impact of the Covid-19 pandemic on families of patients with neuromuscular and neurological disorders | 4 months
  Evaluation of semi-structured questionnaires using thematic analysis
Qualitative evaluation of concerns regarding medical care from the perspective of patients with NMDs and their families during the Covid-19 pandemic | 4 months
  Evaluation of semi-structured questionnaires using thematic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Anita Simonds, MBBS, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spurr L, Tan HL, Wakeman R, Chatwin M, Hughes Z, Simonds A. Psychosocial impact of the COVID-19 pandemic and shielding in adults and children with early-onset neuromuscular and neurological disorders and their families: a mixed-methods study. BMJ Open. 2022 Mar 30;12(3):e055430. doi: 10.1136/bmjopen-2021-055430. PMID 35354630